CLINICAL TRIAL: NCT01995201
Title: A Phase IIIb Study to Evaluate the Efficacy, Safety and Tolerability of Subcutaneous (SC) Tocilizumab (TCZ) Given as Monotherapy or in Combination With Methotrexate (MTX) or Other Non Biologics DMARDs in Subjects With Rheumatoid Arthritis
Brief Title: A Study of Subcutaneous RoActemra/Actemra (Tocilizumab) as Monotherapy or in Combination With Methotrexate or Other Non-Biologic DMARDs in Patients With Active Rheumatoid Arthritis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ML28709; 2013-002429-52 (EudraCT Number)
Record Dates: First submitted 2013-11-01; First posted 2013-11-26 (Estimated); Results first posted 2018-01-26 (Actual); Last update posted 2018-01-26 (Actual); Status verified 2017-06

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Antirheumatic Agents; Methotrexate; tocilizumab

ARMS (3):
- Part 1: All patients (Experimental)
  Interventions: Drug: DMARD; Drug: methotrexate; Drug: tocilizumab [RoActemra/Actemra]
- Part 2 A: Sustained clinical remission (Experimental)
  Interventions: Drug: DMARD; Drug: methotrexate; Drug: tocilizumab [RoActemra/Actemra]
- Part 2 B: Low disease activity (Experimental)
  Interventions: Drug: DMARD; Drug: methotrexate; Drug: tocilizumab [RoActemra/Actemra]

INTERVENTIONS:
Drug: DMARD — non-biological disease-modifying antirheumatic drugs at stable dose
Drug: methotrexate — stable dose
Drug: tocilizumab [RoActemra/Actemra] — 162 mg subcutaneously (SC) qw, Weeks 1-24
  Arms: Part 1: All patients
Drug: tocilizumab [RoActemra/Actemra] — 162 mg SC qw or q2w, Weeks 24-48
  Arms: Part 2 A: Sustained clinical remission
Drug: tocilizumab [RoActemra/Actemra] — 162 mg SC qw, Weeks 24-48
  Arms: Part 2 B: Low disease activity

SUMMARY:
This multicenter, open-label study will evaluate the efficacy and safety of subcutaneously administered RoActemra/Actemra (tocilizumab) as monotherapy or in combination with methotrexate or other non-biologic DMARDs in patients with active rheumatoid arthritis and an inadequate response to non-biologic DMARDs or to one anti-TNF. In Phase 1, all patients will receive RoActemra/Actemra 162 mg subcutaneously (sc) weekly for Weeks 1 to 24, with or without methotrexate or other non-biologic DMARDs. For Part 2, patients who achieve sustained clinical DAS28-ESR remission at Weeks 20 and 24 will be randomized to receive RoActemra/Actemra 162 mg sc either weekly or every 2 weeks for Weeks 24 to 48, with or without methotrexate or other non-biologic DMARDs. Patients who do not achieve sustained clinical remission but achieve low disease activity (DAS-ESR </= 3.2) will continue the initial treatment of RoActemra/Actemra 162 mg sc weekly for Weeks 24 to 48, with or without methotrexate or other non-biologic DMARDs.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients, >/= 18 years of age
* Active rheumatoid arthritis (DAS28-ESR > 3.2), according to the revised (1987) ACR criteria or EULAR/ACR (2010) criteria of > 6 months duration
* Patients with intolerance or inadequate response to methotrexate or other non-biologic DMRADs or inadequate response to a first ant-TNF agent
* Oral corticosteroids (</= 10 mg/day prednisone or equivalent) and non-steroidal anti-inflammatory drugs (NSAIDs; up to the maximum recommended dose) are permitted if on a stable dose regimen for >/= 4 weeks prior to baseline
* Permitted non-biologic DMRAD is allowed if at stable dose for at least 4 weeks prior to baseline
* Females of childbearing potential and males with female partners of childbearing potential must be using a reliable means of contraception as defined by protocol during the study and for at least 3 months following the last dose of RoActemra/Actemra
* Patients with intolerance or inadequate response to methotrexate or other non-biologic DMARDs or inadequate response to first anti-TNF agent

Exclusion Criteria:

* Major surgery (including joint surgery) within 8 weeks prior to screening or planned major surgery within 6 months following baseline
* Rheumatic autoimmune disease other than RA or significant systemic involvement secondary to RA; secondary Sjögren's syndrome with RA is permitted
* Functional Class IV as defined by the ACR Classification of Functional Status in Rheumatoid Arthritis
* Diagnosis of juvenile idiopathic arthritis or juvenile RA and/or RA before the age of 16
* Prior history of current inflammatory joint disease other than RA
* Exposure to tocilizumab (either intravenous [IV] or SC) at any time prior to baseline
* Treatment with any investigational agent with four weeks (or five-half lives of the investigational drug, whichever is longer) of screening
* Intra-articular or parenteral corticosteroids within 4 weeks prior to baseline
* Previous treatment with Abatacept
* History of severe allergic of anaphylactic reactions to human, humanized, or murine monoclonal antibodies
* Evidence of serious uncontrolled concomitant cardiovascular, nervous system, pulmonary, renal, hepatic, endocrine, or gastrointestinal (GI) disease
* History of diverticulitis, diverticulitis requiring antibiotic treatment, or chronic ulcerative lower GI disease such as Crohn's disease, ulcerative colitis, or other symptomatic lower GI conditions that might predispose to perforation
* Known active current or history of recurrent bacterial, viral, fungal, mycobacterial, or other infections (including but not limited to tuberculosis [TB] and atypical mycobacterial disease, hepatitis B and C, and herpes zoster, but excluding fungal infections or nail beds)
* Any major episode of infection requiring hospitalization or treatment with IV antibiotics within 4 weeks of screening or oral antibiotics within 2 weeks of screening
* Active TB requiring treatment within the previous 3 years
* Positive hepatitis B or hepatitis C
* Primary or secondary immunodeficiency (history of or currently active)
* Evidence of active malignant disease, malignancies diagnosed with the previous 10 years (including hematological malignancies and solid tumors, except basal of squamous cell carcinoma of the skin diagnosed within the previous 20 years
* Pregnant and lactating women
* History of alcohol, drug, or chemical abuse within 1 year prior to screening
* Neuropathies or other conditions that might interfere with pain evaluation
* Inadequate hematological, real of liver function

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 401 (Actual)
Dates: Start 2013-09; Primary Completion 2015-07 (Actual); Study Completion 2016-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (41):
- Ireland (5):
  - Co Leitrim
  - Cork
  - Dublin
  - Limerick
  - Waterford
- Portugal (4):
  - Almada
  - Amadora
  - Lisbon
  - Porto
- Spain (32):
  - Elche, Alicante
  - Mérida, Badajoz
  - Palma de Mallorca, Balearic Islands
  - Sabadell, Barcelona
  - Sant Joan Despí, Barcelona
  - Terrassa, Barcelona
  - Jerez de la Frontera, Cadiz
  - Torrelavega, Cantabria
  - Donostia / San Sebastian, Guipuzcoa
  - A Coruña, La Coruña
  - Santiago de Compostela, La Coruña
  - Las Palmas de Gran Canaria, Las Palmas
  - Fuenlabrada, Madrid
  - Cartagena, Murcia
  - El Palmar, Murcia
  - Santa Cruz de Tenerife, Tenerife
  - Valenica, Valencia
  - Bilbao, Vizcaya
  - Alicante
  - Barcelona
  - Burgos
  - Córdoba
  - Granada
  - Guadalajara
  - Madrid
  - Málaga
  - Salamanca
  - Seville
  - Tarragona
  - Toledo
  - Valencia
  - Zaragoza

REFERENCES:
- [Derived] Sanmarti R, Veale DJ, Martin-Mola E, Escudero-Contreras A, Gonzalez C, Ercole L, Alonso R, Fonseca JE; ToSpace Study Group. Reducing or Maintaining the Dose of Subcutaneous Tocilizumab in Patients With Rheumatoid Arthritis in Clinical Remission: A Randomized, Open-Label Trial. Arthritis Rheumatol. 2019 Oct;71(10):1616-1625. doi: 10.1002/art.40905. Epub 2019 Sep 24. PMID 31087542
- [Derived] Choy E, Caporali R, Xavier R, Fautrel B, Sanmarti R, Bao M, Devenport J, Petho-Schramm A. Effects of concomitant glucocorticoids in TOZURA, a common-framework study programme of subcutaneous tocilizumab in rheumatoid arthritis. Rheumatology (Oxford). 2019 Jun 1;58(6):1056-1064. doi: 10.1093/rheumatology/key393. PMID 30649524
- [Derived] Choy E, Caporali R, Xavier R, Fautrel B, Sanmarti R, Bao M, Bernasconi C, Petho-Schramm A. Subcutaneous tocilizumab in rheumatoid arthritis: findings from the common-framework phase 4 study programme TOZURA conducted in 22 countries. Rheumatology (Oxford). 2018 Mar 1;57(3):499-507. doi: 10.1093/rheumatology/kex443. PMID 29244149

RESULTS

PARTICIPANT FLOW:
Groups:
- Phase 1: Tocilizumab Monotherapy: Participants received Tocilizumab (TCZ), 162mg, by sub-cutaneous injection as a single fixed dose monotherapy once a week for 24 weeks.
- Phase 1: Combination Therapy: Participants received Tocilizumab (TCZ), 162mg, by sub-cutaneous injection in combination with oral or sub-cutaneous methotrexate (MTX) or other non-biologic Disease Modifying Anti Rheumatic Drugs (nbDMARDs) once a week for 24 weeks.
- Phase 2 Arm A1: TCZ +/- nbDMARD Once Per Week (qw): Participants who achieved sustained clinical remission (DAS28-ESR <2.6) at Week 20 and Week 24 in Part 1 were randomized to tocilizumab given every week monotherapy or in combination with methotrexate or other non-biologics DMARDs from Week 24 to Week 48.
- Phase 2 Arm A2: TCZ +/- nbDMARD Every Two Weeks (q2w): Participants who achieved sustained clinical remission (DAS28-ESR <2.6) at Week 20 and Week 24 in Part 1 were randomized to tocilizumab given every 2 weeks monotherapy or in combination with methotrexate or other non-biologics DMARDs from Week 24 to Week 48.
- Phase 2 Arm B: Participants With Low Disease Activity: Participants who did not achieve sustained clinical remission at Week 20 and Week 24 but achieve low disease activity (DAS 28-ESR ≤ 3.2) at Week 24 continued with initial treatment of tocilizumab as a single fixed dose monotherapy or in combination with methotrexate or other non-biologics DMARDs from Week 24 to Week 48.
- Phase 2 Arm C: Moderate EULAR Response at Week 24: Patients who achieved moderate EULAR response at Week 24 continued in the study with initial treatment as per investigator's judgement.
- Phase 2 Arm D: Non Responders: Non responders, safety population.
Period: From Baseline Until Week 24
Arm/Group | Phase 1: Tocilizumab Monotherapy | Phase 1: Combination Therapy | Phase 2 Arm A1: TCZ +/- nbDMARD Once Per Week (qw) | Phase 2 Arm A2: TCZ +/- nbDMARD Every Two Weeks (q2w) | Phase 2 Arm B: Participants With Low Disease Activity | Phase 2 Arm C: Moderate EULAR Response at Week 24 | Phase 2 Arm D: Non Responders
Started | 74 | 327 | 0 | 0 | 0 | 0 | 0
Completed | 64 | 281 | 0 | 0 | 0 | 0 | 0
Not Completed | 10 | 46 | 0 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 4 | 15 | 0 | 0 | 0 | 0 | 0
Not completed — Anaphylaxis or hypersensitivity reaction | 0 | 3 | 0 | 0 | 0 | 0 | 0
Not completed — Death | 0 | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Lack of Efficacy | 2 | 5 | 0 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 2 | 3 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 2 | 8 | 0 | 0 | 0 | 0 | 0
Not completed — Physician Decision | 0 | 2 | 0 | 0 | 0 | 0 | 0
Not completed — Protocol Violation | 0 | 9 | 0 | 0 | 0 | 0 | 0
Period: From Week 24 Until Week 48
Arm/Group | Phase 1: Tocilizumab Monotherapy | Phase 1: Combination Therapy | Phase 2 Arm A1: TCZ +/- nbDMARD Once Per Week (qw) | Phase 2 Arm A2: TCZ +/- nbDMARD Every Two Weeks (q2w) | Phase 2 Arm B: Participants With Low Disease Activity | Phase 2 Arm C: Moderate EULAR Response at Week 24 | Phase 2 Arm D: Non Responders
Started | 0 | 0 | 89 | 90 | 95 | 67 | 2
Completed | 0 | 0 | 84 | 89 | 89 | 59 | 0
Not Completed | 0 | 0 | 5 | 1 | 6 | 8 | 2
Not completed — Adverse Event | 0 | 0 | 2 | 1 | 1 | 3 | 1
Not completed — Death | 0 | 0 | 0 | 0 | 0 | 2 | 0
Not completed — Lack of Efficacy | 0 | 0 | 1 | 0 | 0 | 2 | 1
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 1 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 1 | 0 | 1 | 0 | 0
Not completed — Physician Decision | 0 | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Protocol Violation | 0 | 0 | 1 | 0 | 2 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Phase 1: Tocilizumab Monotherapy | Phase 1: Combination Therapy | Total
Number analyzed (Participants) | 74 | 327 | 401
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.5 (12.7) | 53.6 (12.2) | 53.6 (12.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 62 | 264 | 326
  Male | 12 | 63 | 75

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Achieving Sustained Clinical Remission, Disease Activity Scale 28 - Erythrocyte Sedimentation Rate <26 (DAS28-ESR <2.6) at Week 20 and Week 24
Description: The DAS 28 is a combined index for measuring disease activity in RA. The index includes the assessment of 28 joints for swelling and tenderness, acute phase response (ESR or CRP) and general health status. For this study ESR was used to calculate the DAS 28 score.
Time Frame: Week 20 and Week 24
Population: Analyses were conducted on the Full Analysis Set (FAS), i.e. all patients included in the study who received at least one dose of SC TCZ.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Phase 1: Tocilizumab Monotherapy | Phase 1: Combination Therapy
Number analyzed (Participants) | 74 | 327
Percentage of participants | 48.4 [35.75 to 61.27] | 52.9 [46.83 to 58.83]
Statistical Analysis 1: Comparison: Phase 1: Tocilizumab Monotherapy vs Phase 1: Combination Therapy; Test type: Other; p = 0.5231, Chi-squared

2. Secondary Outcome: Mean Change in Disease Activity Score 28 - Erythrocyte Sedimentation Rate(DAS28-ESR)
Description: as for outcome 1
Time Frame: From week 24 up to week 48
Population: Analysis was conducted on the FAS
Measure: Mean (Standard Deviation); unit: mm/hr
Groups:
- Phase 2 Arm A1: TCZ +/- nbDMARD Once Per Week (qw): Participants who achieve sustained clinical remission (DAS28-ESR <2.6) at Week 20 and Week 24 in Part 1 were randomized to tocilizumab given every week monotherapy or in combination with methotrexate or other non-biologics DMARDs from Week 24 to Week 48.
- Phase 2 Arm A2: TCZ +/- nbDMARD Every Two Weeks (q2w): Participants who achieve sustained clinical remission (DAS28-ESR <2.6) at Week 20 and Week 24 in Part 1 will be randomized to tocilizumab given every 2 weeks monotherapy or in combination with methotrexate or other non-biologics DMARDs from Week 24 to Week 48.
Arm/Group | Phase 2 Arm A1: TCZ +/- nbDMARD Once Per Week (qw) | Phase 2 Arm A2: TCZ +/- nbDMARD Every Two Weeks (q2w)
Number analyzed (Participants) | 89 | 90
mm/hr
  Week 24 | -4.07 (1.03) | -4.01 (1.13)
  Week 28: number analyzed (Participants) | 87 | 88
  Week 28 | -3.94 (1.22) | -3.78 (1.31)
  Week 32: number analyzed (Participants) | 86 | 90
  Week 32 | -3.97 (1.38) | -3.77 (1.17)
  Week 36: number analyzed (Participants) | 86 | 88
  Week 36 | -3.82 (1.53) | -3.90 (1.16)
  Week 40: number analyzed (Participants) | 84 | 88
  Week 40 | -3.95 (1.26) | -3.84 (1.19)
  Week 44: number analyzed (Participants) | 82 | 88
  Week 44 | -4.05 (1.17) | -3.76 (1.17)
  Week 48: number analyzed (Participants) | 82 | 88
  Week 48 | -4.14 (1.24) | -3.68 (1.32)

3. Secondary Outcome: Percentage of Patients Allocated in Groups A1 and A2 Who Remain With Clinical Remission Activity (DAS 28 ESR <2.6) up to Week 48
Description: The DAS28 is a combined index for measuring disease activity in RA. The index includes the assessment of 28 joints for swelling and tenderness, acute phase response (ESR or CRP), and general health status. For this study ESR will be used to calculate the DAS28 score.
Time Frame: From week 28 up to week 48
Population: Analysis was conducted on the FAS
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Phase 2 Arm A1: TCZ +/- nbDMARD Once Per Week (qw) | Phase 2 Arm A2: TCZ +/- nbDMARD Every Two Weeks (q2w)
Number analyzed (Participants) | 89 | 90
Percentage of participants
  Week 28 | 88.5 [79.88 to 94.35] | 84.1 [74.75 to 91.02]
  Week 32: number analyzed (Participants) | 87 | 90
  Week 32 | 87.2 [78.27 to 93.44] | 81.1 [71.49 to 88.59]
  Week 36: number analyzed (Participants) | 86 | 89
  Week 36 | 80.2 [70.25 to 88.04] | 86.4 [77.39 to 92.75]
  Week 40: number analyzed (Participants) | 84 | 88
  Week 40 | 82.1 [72.26 to 89.65] | 80.7 [70.88 to 88.32]
  Week 44: number analyzed (Participants) | 82 | 89
  Week 44 | 89.0 [80.18 to 94.86] | 78.4 [68.35 to 86.47]
  Week 48: number analyzed (Participants) | 84 | 89
  Week 48 | 91.5 [83.20 to 96.50] | 73.9 [63.41 to 82.66]

4. Secondary Outcome: Percentage of Patients Reporting Change in DAS 28 ESR >1.2 Until Week 48
Description: as for outcome 3
Time Frame: From week 28 up to week 48
Population: Analysis was conducted on the FAS
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Phase 2 Arm A1: TCZ +/- nbDMARD Once Per Week (qw) | Phase 2 Arm A2: TCZ +/- nbDMARD Every Two Weeks (q2w)
Number analyzed (Participants) | 89 | 90
Percentage of participants
  Week 28: number analyzed (Participants) | 88 | 90
  Week 28 | 96.6 [90.25 to 99.28] | 96.6 [90.36 to 99.29]
  Week 32: number analyzed (Participants) | 87 | 90
  Week 32 | 96.5 [90.14 to 99.27] | 95.6 [89.01 to 98.78]
  Week 36: number analyzed (Participants) | 86 | 89
  Week 36 | 93.0 [85.43 to 97.40] | 97.7 [92.03 to 99.72]
  Week 40: number analyzed (Participants) | 84 | 88
  Week 40 | 98.8 [93.54 to 99.97] | 98.9 [93.83 to 99.97]
  Week 44: number analyzed (Participants) | 82 | 89
  Week 44 | 98.8 [93.39 to 99.97] | 95.5 [88.77 to 98.75]
  Week 48: number analyzed (Participants) | 84 | 89
  Week 48 | 100.0 [NA to NA] — NA because the central value is 100% | 95.5 [88.77 to 98.75]

5. Secondary Outcome: Percentage of Patients With American College of Rheumatology (ACR20, 50, 70, 90) Response Scores Until Week 24
Description: The definition of improvement of ACR core set of outcome measures includes an improvement equal or higher to the 20%, 50%, 70%, 90% compared to Baseline in both Swollen Joint Count (SJC) and Tender Joint Count (TJC) as well as in three out of five additional parameters: Physician's Global Assessment of disease activity VAS, patient's Global Assessment of disease activity VAS, patient's assessment of pain VAS, HAQ-DI, and acute phase reactant (either CRP or erythrocyte sedimentation rate [ESR]).
Time Frame: From week 2 until week 24
Population: Analysis was conducted on the FAS
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Phase 1: Tocilizumab Monotherapy | Phase 1: Combination Therapy
Number analyzed (Participants) | 74 | 327
Percentage of participants
  ACR20 - Week 2: number analyzed (Participants) | 74 | 319
  ACR20 - Week 2 | 27.0 [17.35 to 38.61] | 31.7 [26.59 to 37.08]
  ACR20 - Week 4: number analyzed (Participants) | 73 | 312
  ACR20 - Week 4 | 50.7 [38.72 to 62.60] | 49.7 [44.00 to 55.37]
  ACR20 - Week 8: number analyzed (Participants) | 73 | 300
  ACR20 - Week 8 | 67.1 [55.13 to 77.67] | 67.0 [61.36 to 72.30]
  ACR20 - Week 12: number analyzed (Participants) | 70 | 296
  ACR20 - Week 12 | 80.0 [68.73 to 88.61] | 74.7 [69.31 to 79.52]
  ACR20 - Week 16: number analyzed (Participants) | 69 | 292
  ACR20 - Week 16 | 79.7 [68.31 to 88.44] | 75.7 [70.35 to 80.49]
  ACR20 - Week 20: number analyzed (Participants) | 65 | 284
  ACR20 - Week 20 | 73.8 [61.46 to 83.97] | 81.0 [75.93 to 85.38]
  ACR20 - Week 24: number analyzed (Participants) | 64 | 281
  ACR20 - Week 24 | 79.7 [67.77 to 88.72] | 83.3 [78.39 to 87.44]
  ACR20 - LOCF visit: number analyzed (Participants) | 74 | 319
  ACR20 - LOCF visit | 77.0 [67.77 to 88.72] | 79.0 [78.39 to 87.44]
  ACR50 - week 2: number analyzed (Participants) | 74 | 319
  ACR50 - week 2 | 9.5 [3.89 to 18.52] | 13.2 [9.66 to 17.38]
  ACR50 - week 4: number analyzed (Participants) | 73 | 312
  ACR50 - week 4 | 20.5 [11.98 to 31.62] | 25.3 [20.59 to 30.53]
  ACR50 - week 8: number analyzed (Participants) | 73 | 300
  ACR50 - week 8 | 37.0 [25.97 to 49.09] | 41.3 [35.70 to 47.14]
  ACR50 - week 12: number analyzed (Participants) | 70 | 296
  ACR50 - week 12 | 51.4 [39.17 to 63.56] | 52.7 [46.84 to 58.51]
  ACR50 - week 16: number analyzed (Participants) | 69 | 292
  ACR50 - week 16 | 53.6 [41.20 to 65.72] | 52.4 [46.50 to 58.25]
  ACR50 - week 20: number analyzed (Participants) | 65 | 284
  ACR50 - week 20 | 58.5 [45.56 to 70.56] | 58.5 [52.48 to 64.24]
  ACR50 - week 24: number analyzed (Participants) | 64 | 281
  ACR50 - week 24 | 59.4 [46.37 to 71.49] | 58.7 [52.72 to 64.53]
  ACR50 - LOCF visit: number analyzed (Participants) | 74 | 319
  ACR50 - LOCF visit | 55.4 [46.37 to 71.49] | 54.2 [52.72 to 64.53]
  ACR70 - week 2: number analyzed (Participants) | 74 | 319
  ACR70 - week 2 | 5.4 [1.49 to 13.27] | 2.8 [1.30 to 5.29]
  ACR70 - week 4: number analyzed (Participants) | 73 | 312
  ACR70 - week 4 | 12.3 [5.80 to 22.12] | 10.6 [7.39 to 14.53]
  ACR70 - week 8: number analyzed (Participants) | 73 | 300
  ACR70 - week 8 | 17.8 [9.84 to 28.53] | 22.7 [18.05 to 27.83]
  ACR70 - week 12: number analyzed (Participants) | 70 | 296
  ACR70 - week 12 | 32.9 [22.09 to 45.12] | 27.0 [22.05 to 32.47]
  ACR70 - week 16: number analyzed (Participants) | 69 | 292
  ACR70 - week 16 | 29.0 [18.69 to 41.16] | 32.2 [26.87 to 37.88]
  ACR70 - week 20: number analyzed (Participants) | 65 | 284
  ACR70 - week 20 | 33.8 [22.57 to 46.65] | 36.6 [31.01 to 42.52]
  ACR70 - week 24: number analyzed (Participants) | 64 | 281
  ACR70 - week 24 | 40.6 [28.51 to 53.63] | 37.7 [32.03 to 43.67]
  ACR70 - LOCF visit: number analyzed (Participants) | 74 | 319
  ACR70 - LOCF visit | 37.8 [28.51 to 53.63] | 33.9 [32.03 to 43.67]
  ACR90 - week 2: number analyzed (Participants) | 74 | 319
  ACR90 - week 2 | 1.4 [0.03 to 7.30] | 0.9 [0.19 to 2.72]
  ACR90 - week 4: number analyzed (Participants) | 73 | 312
  ACR90 - week 4 | 2.7 [0.33 to 9.55] | 1.6 [0.52 to 3.70]
  ACR90 - week 8: number analyzed (Participants) | 73 | 300
  ACR90 - week 8 | 6.8 [2.26 to 15.26] | 7.3 [4.65 to 10.89]
  ACR90 - week 12: number analyzed (Participants) | 70 | 296
  ACR90 - week 12 | 12.9 [6.05 to 23.01] | 8.8 [5.82 to 12.61]
  ACR90 - week 16: number analyzed (Participants) | 69 | 292
  ACR90 - week 16 | 13.0 [6.14 to 23.32] | 12.0 [8.49 to 16.27]
  ACR90 - week 20: number analyzed (Participants) | 65 | 284
  ACR90 - week 20 | 13.8 [6.53 to 24.66] | 13.7 [9.95 to 18.29]
  ACR90 - week 24: number analyzed (Participants) | 64 | 281
  ACR90 - week 24 | 23.4 [13.75 to 35.69] | 16.7 [12.56 to 21.61]
  ACR90 - LOCF visit: number analyzed (Participants) | 74 | 319
  ACR90 - LOCF visit | 20.3 [13.75 to 35.69] | 15.0 [12.56 to 21.61]

6. Secondary Outcome: Percentage of Patients With American College of Rheumatology (ACR20, 50, 70, 90) Response Scores Until Week 48
Description: as for outcome 5
Time Frame: From week 28 until week 48
Population: Analysis was conducted on the FAS
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Phase 2 Arm A1: TCZ +/- nbDMARD Once Per Week (qw) | Phase 2 Arm A2: TCZ +/- nbDMARD Every Two Weeks (q2w)
Number analyzed (Participants) | 89 | 90
Percentage of participants
  ACR20 - Week 28: number analyzed (Participants) | 88 | 90
  ACR20 - Week 28 | 90.0 [82.7 to 95.99] | 92.2 [84.63 to 96.82]
  ACR20 - Week 32: number analyzed (Participants) | 87 | 90
  ACR20 - Week 32 | 93.1 [85.59 to 97.43] | 94.4 [87.51 to 98.17]
  ACR20 - Week 36: number analyzed (Participants) | 86 | 89
  ACR20 - Week 36 | 84.9 [75.54 to 91.70] | 91.0 [83.05 to 96.04]
  ACR20 - Week 40: number analyzed (Participants) | 84 | 88
  ACR20 - Week 40 | 88.1 [79.19 to 94.14] | 93.2 [85.75 to 97.46]
  ACR20 - Week 44: number analyzed (Participants) | 82 | 89
  ACR20 - Week 44 | 91.5 [83.20 to 96.50] | 91.0 [83.05 to 96.04]
  ACR20 - Week 48: number analyzed (Participants) | 84 | 89
  ACR20 - Week 48 | 96.4 [89.92 to 99.26] | 88.8 [80.31 to 94.48]
  ACR20 - LOCF visit | 95.5 [88.89 to 98.76] | 87.8 [79.18 to 93.74]
  ACR50 - Week 28: number analyzed (Participants) | 88 | 90
  ACR50 - Week 28 | 79.5 [69.61 to 87.40] | 81.1 [71.49 to 88.59]
  ACR50 - Week 32: number analyzed (Participants) | 87 | 90
  ACR50 - Week 32 | 85.1 [75.80 to 91.80] | 83.3 [74.00 to 90.36]
  ACR50 - Week 36: number analyzed (Participants) | 86 | 89
  ACR50 - Week 36 | 74.4 [63.87 to 83.22] | 83.1 [73.73 to 90.25]
  ACR50 - Week 40: number analyzed (Participants) | 84 | 88
  ACR50 - Week 40 | 79.8 [69.59 to 87.75] | 81.8 [72.16 to 89.24]
  ACR50 - Week 44: number analyzed (Participants) | 82 | 89
  ACR50 - Week 44 | 80.5 [70.26 to 88.42] | 78.7 [68.69 to 86.63]
  ACR50 - Week 48: number analyzed (Participants) | 84 | 89
  ACR50 - Week 48 | 88.1 [79.19 to 94.14] | 79.8 [69.93 to 87.55]
  ACR50 - LOCF visit | 84.3 [75.02 to 91.12] | 78.9 [69.01 to 86.79]
  ACR70 - Week 28: number analyzed (Participants) | 88 | 90
  ACR70 - Week 28 | 59.1 [48.09 to 69.46] | 57.8 [46.91 to 68.12]
  ACR70 - Week 32: number analyzed (Participants) | 87 | 90
  ACR70 - Week 32 | 65.5 [54.56 to 75.39] | 54.4 [43.60 to 64.98]
  ACR70 - Week 36: number analyzed (Participants) | 86 | 89
  ACR70 - Week 36 | 61.6 [50.51 to 71.92] | 62.9 [52.03 to 72.93]
  ACR70 - Week 40: number analyzed (Participants) | 84 | 88
  ACR70 - Week 40 | 65.5 [54.31 to 75.52] | 59.1 [48.09 to 69.46]
  ACR70 - Week 44: number analyzed (Participants) | 82 | 89
  ACR70 - Week 44 | 67.1 [55.81 to 77.06] | 59.6 [48.62 to 69.83]
  ACR70 - Week 48: number analyzed (Participants) | 84 | 89
  ACR70 - Week 48 | 71.4 [60.53 to 80.76] | 65.2 [54.33 to 74.96]
  ACR70 - LOCF visit | 68.5 [57.83 to 77.97] | 64.4 [53.65 to 74.26]
  ACR90 - Week 28: number analyzed (Participants) | 88 | 90
  ACR90 - Week 28 | 27.3 [18.32 to 37.81] | 32.2 [22.75 to 42.90]
  ACR90 - Week 32: number analyzed (Participants) | 87 | 90
  ACR90 - Week 32 | 35.6 [25.65 to 46.62] | 31.1 [21.77 to 41.74]
  ACR90 - Week 36: number analyzed (Participants) | 86 | 89
  ACR90 - Week 36 | 33.7 [23.88 to 44.72] | 30.3 [21.03 to 40.99]
  ACR90 - Week 40: number analyzed (Participants) | 84 | 88
  ACR90 - Week 40 | 41.7 [31.00 to 52.94] | 29.5 [20.29 to 40.22]
  ACR90 - Week 44: number analyzed (Participants) | 82 | 89
  ACR90 - Week 44 | 34.1 [24.03 to 45.45] | 27.0 [18.10 to 37.42]
  ACR90 - Week 48: number analyzed (Participants) | 84 | 89
  ACR90 - Week 48 | 45.2 [34.34 to 56.48] | 32.6 [23.02 to 43.34]
  ACR90 - LOCF visit | 42.7 [32.26 to 53.63] | 32.2 [22.75 to 42.90]

7. Secondary Outcome: Number of Patients With Good and Moderate Clinical Response According to European League Against Rheumatism (EULAR) Response Scores up to Week 24
Description: DAS28-based EULAR response criteria were used to measure individual response as good or moderate depending on the extent of change from baseline and the level of disease activity reached. Good responders: change from baseline >1.2 with DAS28 ≤3.2; moderate responders: change from baseline >1.2 with DAS28 >3.2 to ≤5.1 or change from baseline >0.6 to =<1.2 with DAS28 ≤5.1.
Time Frame: From week 2 until week 24
Population: Analysis was conducted on the FAS
Measure: Number; unit: Number of participants
Arm/Group | Phase 1: Tocilizumab Monotherapy | Phase 1: Combination Therapy
Number analyzed (Participants) | 74 | 327
Number of participants
  Good response - week 2: number analyzed (Participants) | 74 | 319
  Good response - week 2 | 14 | 61
  Moderate response - week 2: number analyzed (Participants) | 74 | 319
  Moderate response - week 2 | 36 | 196
  Good response - week 4: number analyzed (Participants) | 73 | 312
  Good response - week 4 | 18 | 109
  Moderate response - week 4: number analyzed (Participants) | 73 | 312
  Moderate response - week 4 | 49 | 175
  Good response - week 8: number analyzed (Participants) | 73 | 300
  Good response - week 8 | 37 | 162
  Moderate response - week 8: number analyzed (Participants) | 73 | 300
  Moderate response - week 8 | 32 | 121
  Good response - week 12: number analyzed (Participants) | 70 | 296
  Good response - week 12 | 41 | 194
  Moderate response - week 12: number analyzed (Participants) | 70 | 296
  Moderate response - week 12 | 27 | 95
  Good response - week 16: number analyzed (Participants) | 69 | 292
  Good response - week 16 | 45 | 209
  Moderate response - week 16: number analyzed (Participants) | 69 | 292
  Moderate response - week 16 | 22 | 76
  Good response - week 20: number analyzed (Participants) | 65 | 284
  Good response - week 20 | 45 | 221
  Moderate response - week 20: number analyzed (Participants) | 65 | 284
  Moderate response - week 20 | 18 | 56
  Good response - week 24: number analyzed (Participants) | 64 | 281
  Good response - week 24 | 48 | 225
  Moderate response - week 24: number analyzed (Participants) | 64 | 281
  Moderate response - week 24 | 16 | 53
  Good response - LOCF visit | 54 | 247
  Moderate response - LOCF visit | 19 | 73

8. Secondary Outcome: Number of Patients With Clinical Response According to European League Against Rheumatism (EULAR) Response Scores up to Week 48
Description: as for outcome 7
Time Frame: From week 28 until week 48
Population: Analysis was conducted on the FAS.
Measure: Number; unit: Number of participants
Arm/Group | Phase 2 Arm A1: TCZ +/- nbDMARD Once Per Week (qw) | Phase 2 Arm A2: TCZ +/- nbDMARD Every Two Weeks (q2w)
Number analyzed (Participants) | 89 | 90
Number of participants
  Good response - week 28: number analyzed (Participants) | 88 | 90
  Good response - week 28 | 82 | 77
  Moderate response - week 28: number analyzed (Participants) | 88 | 90
  Moderate response - week 28 | 5 | 10
  Good response - week 32: number analyzed (Participants) | 87 | 90
  Good response - week 32 | 79 | 81
  Moderate response - week 32: number analyzed (Participants) | 87 | 90
  Moderate response - week 32 | 6 | 9
  Good response - week 36: number analyzed (Participants) | 86 | 89
  Good response - week 36 | 75 | 80
  Moderate response - week 36: number analyzed (Participants) | 86 | 89
  Moderate response - week 36 | 9 | 8
  Good response - week 40: number analyzed (Participants) | 84 | 88
  Good response - week 40 | 75 | 81
  Moderate response - week 40: number analyzed (Participants) | 84 | 88
  Moderate response - week 40 | 9 | 7
  Good response - week 44: number analyzed (Participants) | 82 | 89
  Good response - week 44 | 78 | 75
  Moderate response - week 44: number analyzed (Participants) | 82 | 89
  Moderate response - week 44 | 4 | 13
  Good response - week 48: number analyzed (Participants) | 84 | 89
  Good response - week 48 | 78 | 73
  Moderate response - week 48: number analyzed (Participants) | 84 | 89
  Moderate response - week 48 | 4 | 15
  Good response - LOCF visit | 84 | 74
  Moderate response - LOCF visit | 5 | 16

9. Secondary Outcome: Mean Change in Clinical Disease Activity Index (CDAI) From Baseline up to Week 24
Description: Clinical Disease Activity Index (CDAI) is an index for measuring disease activity in rheumatoid arthritis (RA). The index was calculated using the following formula: CDAI = number of swollen joints using the 28-joint count (SJC28) + number of tender joints using the 28-joint count (TJC28) + patient global assessment of disease (PGA) based on 10 centimeter [cm] Visual Analog Scale [VAS] + physician global assessment of disease (PhGA) based on 10 cm VAS. VAS assessments involved a 10 cm horizontal scale from 0 (no disease activity) to 10 (maximum disease activity). Total CDAI scores ranged from 0 to 76, with higher scores indicating increased disease activity. A negative change from baseline indicates an improvement.
Time Frame: From baseline to Week 24
Population: Analysis was conducted on the FAS.
Measure: Mean (Standard Deviation); unit: CDAI score
Arm/Group | Phase 1: Tocilizumab Monotherapy | Phase 1: Combination Therapy
Number analyzed (Participants) | 74 | 327
CDAI score
  Baseline values | 33.06 (12.45) | 32.06 (12.28)
  Week 2: number analyzed (Participants) | 74 | 319
  Week 2 | -7.54 (9.57) | -8.62 (9.22)
  Week 4: number analyzed (Participants) | 73 | 312
  Week 4 | -13.03 (10.91) | -13.23 (10.65)
  Week 8: number analyzed (Participants) | 73 | 299
  Week 8 | -18.06 (11.05) | -18.46 (11.61)
  Week 12: number analyzed (Participants) | 70 | 296
  Week 12 | -21.56 (11.77) | -20.60 (11.42)
  Week 16: number analyzed (Participants) | 69 | 290
  Week 16 | -23.01 (12.33) | -21.79 (11.57)
  Week 20: number analyzed (Participants) | 65 | 284
  Week 20 | -24.07 (11.97) | -22.88 (12.10)
  Week 24: number analyzed (Participants) | 64 | 281
  Week 24 | -25.80 (13.31) | -23.43 (11.62)
  LOCF visit | -24.42 (13.50) | -21.58 (12.85)

10. Secondary Outcome: Mean Change From Baseline in Clinical Disease Activity Index (CDAI) up to Week 48
Description: as for outcome 9
Time Frame: From week 24 until week 48
Population: Analysis was conducted on the FAS.
Measure: Mean (Standard Deviation); unit: CDAI score
Arm/Group | Phase 2 Arm A1: TCZ +/- nbDMARD Once Per Week (qw) | Phase 2 Arm A2: TCZ +/- nbDMARD Every Two Weeks (q2w)
Number analyzed (Participants) | 89 | 90
CDAI score
  Baseline values | 29.27 (10.90) | 29.64 (12.13)
  Week 24 | -25.54 (10.60) | -25.34 (12.10)
  Week 28: number analyzed (Participants) | 88 | 89
  Week 28 | -24.75 (10.64) | -24.01 (12.30)
  Week 32: number analyzed (Participants) | 87 | 90
  Week 32 | -24.56 (12.93) | -25.12 (11.64)
  Week 36: number analyzed (Participants) | 86 | 88
  Week 36 | -23.90 (11.56) | -25.45 (11.42)
  Week 40: number analyzed (Participants) | 84 | 88
  Week 40 | -25.16 (10.43) | -25.45 (11.75)
  Week 44: number analyzed (Participants) | 82 | 89
  Week 44 | -25.45 (10.11) | -25.26 (11.75)
  Week 48: number analyzed (Participants) | 83 | 89
  Week 48 | -26.44 (11.13) | -25.13 (12.51)
  LOCF visit | -25.74 (11.29) | -24.87 (12.67)

11. Secondary Outcome: Mean Change in Simplified Disease Activity Index (SDAI) From Baseline up to Week 24
Description: Simplified Disease Activity Index (SDAI) is the numerical sum of five outcome parameters: TJC and SJC (based on a 28-joint assessment), PtGA and PhGA (based on 0-10 cm VAS, where 0 = no disease activity and 10 = worst disease activity), and CRP. SDAI total score ranges from 0 (no disease activity) to 86 (maximal disease activity), where higher scores represents higher disease activity. The SDAI =< 3.3 indicates disease remission, > 3.4 to 11 indicates low disease activity, > 11 to 26 indicates moderate disease activity, and > 26 indicates high disease activity.
Time Frame: From baseline to Week 24
Population: Analysis was conducted on the FAS
Measure: Mean (Standard Deviation); unit: SDAI score
Arm/Group | Phase 1: Tocilizumab Monotherapy | Phase 1: Combination Therapy
Number analyzed (Participants) | 74 | 327
SDAI score
  Baseline values: number analyzed (Participants) | 74 | 324
  Baseline values | 48.66 (31.48) | 44.40 (22.91)
  Week 2: number analyzed (Participants) | 72 | 309
  Week 2 | -20.45 (19.01) | -19.50 (18.75)
  Week 4: number analyzed (Participants) | 70 | 308
  Week 4 | -27.86 (23.54) | -24.34 (20.98)
  Week 8: number analyzed (Participants) | 72 | 292
  Week 8 | -32.61 (26.84) | -29.34 (21.96)
  Week 12: number analyzed (Participants) | 70 | 291
  Week 12 | -36.23 (27.04) | -30.95 (23.58)
  Week 16: number analyzed (Participants) | 69 | 286
  Week 16 | -37.82 (31.09) | -32.66 (22.79)
  Week 20: number analyzed (Participants) | 64 | 277
  Week 20 | -36.79 (25.47) | -33.95 (23.05)
  Week 24: number analyzed (Participants) | 63 | 277
  Week 24 | -41.38 (31.51) | -34.80 (22.44)
  LOCF visit: number analyzed (Participants) | 74 | 324
  LOCF visit | -39.15 (30.45) | -32.73 (22.84)

12. Secondary Outcome: Mean Change in Simplified Disease Activity Index (SDAI) From Week 24 up to Week 48
Description: Simplified Disease Activity Index (SDAI) which is the numerical sum of five outcome parameters: TJC and SJC (based on a 28-joint assessment), PtGA and PhGA (based on 0-10 cm VAS, where 0 = no disease activity and 10 = worst disease activity), and CRP. SDAI total score ranges from 0 (no disease activity) to 86 (maximal disease activity), where higher scores represents higher disease activity. The SDAI =< 3.3 indicates disease remission, > 3.4 to 11 indicates low disease activity, > 11 to 26 indicates moderate disease activity, and > 26 indicates high disease activity.
Time Frame: From week 24 until week 48
Population: Analysis was conducted on the FAS
Measure: Mean (Standard Deviation); unit: SDAI score
Arm/Group | Phase 2 Arm A1: TCZ +/- nbDMARD Once Per Week (qw) | Phase 2 Arm A2: TCZ +/- nbDMARD Every Two Weeks (q2w)
Number analyzed (Participants) | 89 | 90
SDAI score
  Baseline values: number analyzed (Participants) | 89 | 89
  Baseline values | 41.45 (24.90) | 40.92 (21.42)
  Week 24: number analyzed (Participants) | 88 | 90
  Week 24 | -37.02 (24.60) | -35.88 (20.71)
  Week 28: number analyzed (Participants) | 86 | 87
  Week 28 | -35.15 (25.90) | -34.50 (20.66)
  Week 32: number analyzed (Participants) | 86 | 90
  Week 32 | -35.60 (26.97) | -34.88 (20.53)
  Week 36: number analyzed (Participants) | 86 | 88
  Week 36 | -35.29 (26.55) | -35.35 (20.07)
  Week 40: number analyzed (Participants) | 83 | 88
  Week 40 | -37.26 (25.48) | -35.70 (19.80)
  Week 44: number analyzed (Participants) | 82 | 89
  Week 44 | -37.09 (25.17) | -35.06 (21.77)
  Week 48: number analyzed (Participants) | 82 | 88
  Week 48 | -37.93 (26.32) | -35.02 (21.74)
  LOCF visit | -36.93 (25.75) | -34.69 (21.75)

13. Secondary Outcome: Mean Change From Baseline in Total Tender Joint Counts (TJC) Until Week 24
Description: TCJ is a clinical assessment of 68 joints which are classified as tender/not tender by pressure and joint manipulation on physical examination. Joint prosthesis, arthrodesis or fused joints are not be taken into consideration.
Time Frame: From baseline to Week 24
Population: Analysis was conducted on the FAS.
Measure: Mean (Standard Deviation); unit: TJC
Arm/Group | Phase 1: Tocilizumab Monotherapy | Phase 1: Combination Therapy
Number analyzed (Participants) | 74 | 327
TJC
  Baseline visit | 18.05 (12.98) | 19.12 (13.38)
  Week 2: number analyzed (Participants) | 74 | 319
  Week 2 | -4.31 (7.56) | -5.00 (8.06)
  Week 4: number analyzed (Participants) | 73 | 312
  Week 4 | -7.04 (11.77) | -7.96 (9.43)
  Week 8: number analyzed (Participants) | 73 | 300
  Week 8 | -9.81 (10.37) | -10.90 (11.10)
  Week 12: number analyzed (Participants) | 70 | 296
  Week 12 | -12.27 (10.47) | -12.01 (10.88)
  Week 16: number analyzed (Participants) | 69 | 291
  Week 16 | -13.43 (12.35) | -13.09 (11.02)
  Week 20: number analyzed (Participants) | 65 | 284
  Week 20 | -13.65 (11.73) | -13.70 (11.48)
  Week 24: number analyzed (Participants) | 64 | 281
  Week 24 | -15.47 (13.35) | -14.20 (11.46)
  LOCF visit | -14.36 (12.87) | -13.19 (11.75)

14. Secondary Outcome: Mean Change From Baseline in Total Tender Joint Counts (TJC) Until Week 48
Description: as for outcome 13
Time Frame: From week 24 until week 48
Population: Analysis was conducted on the FAS.
Measure: Mean (Standard Deviation); unit: TJC
Arm/Group | Phase 2 Arm A1: TCZ +/- nbDMARD Once Per Week (qw) | Phase 2 Arm A2: TCZ +/- nbDMARD Every Two Weeks (q2w)
Number analyzed (Participants) | 89 | 90
TJC
  Baseline values | 15.42 (9.05) | 15.97 (12.77)
  Week 28: number analyzed (Participants) | 88 | 90
  Week 28 | -13.66 (8.44) | -12.88 (11.52)
  Week 32: number analyzed (Participants) | 87 | 90
  Week 32 | -13.40 (8.99) | -13.88 (11.43)
  Week 36: number analyzed (Participants) | 86 | 89
  Week 36 | -13.13 (8.82) | -13.78 (11.70)
  Week 40: number analyzed (Participants) | 84 | 88
  Week 40 | -14.06 (8.58) | -14.49 (12.07)
  Week 44: number analyzed (Participants) | 82 | 89
  Week 44 | -14.32 (8.25) | -13.93 (11.62)
  Week 48: number analyzed (Participants) | 84 | 89
  Week 48 | -14.40 (8.61) | -13.43 (12.17)
  LOCF visit | -13.96 (8.68) | -13.27 (12.20)

15. Secondary Outcome: Mean Change in Total Swollen Joint Counts (SJC) From Baseline Until Week 24
Description: SJC is a clinical assessment of 66 joints classified as swollen/not swollen by pressure and joint manipulation on physical examination. Joint prosthesis, arthrodesis or fused joints will not be taken into consideration for swelling.
Time Frame: From baseline to Week 24
Population: Analysis was conducted on the FAS.SJC
Measure: Mean (Standard Deviation); unit: SJC
Arm/Group | Phase 1: Tocilizumab Monotherapy | Phase 1: Combination Therapy
Number analyzed (Participants) | 74 | 327
SJC
  Baseline values | 10.05 (7.99) | 9.76 (6.64)
  Week 2: number analyzed (Participants) | 74 | 319
  Week 2 | -3.22 (4.40) | -3.42 (5.10)
  Week 4: number analyzed (Participants) | 73 | 312
  Week 4 | -5.07 (5.58) | -5.46 (5.41)
  Week 8: number analyzed (Participants) | 73 | 300
  Week 8 | -7.38 (6.47) | -6.81 (6.03)
  Week 12: number analyzed (Participants) | 70 | 296
  Week 12 | -7.93 (7.13) | -7.60 (6.00)
  Week 16: number analyzed (Participants) | 69 | 290
  Week 16 | -8.35 (7.71) | -8.01 (6.05)
  Week 20: number analyzed (Participants) | 65 | 284
  Week 20 | -8.72 (7.56) | -8.37 (6.50)
  Week 24: number analyzed (Participants) | 64 | 281
  Week 24 | -9.13 (7.66) | -8.38 (6.59)
  LOCF visit | -8.47 (7.48) | -7.71 (6.67)

16. Secondary Outcome: Mean Change in Total Swollen Joint Counts (SJC) From Baseline Until Week 48
Description: as for outcome 15
Time Frame: From week 24 until week 48
Population: Analysis was conducted on the FAS.
Measure: Mean (Standard Deviation); unit: SJC
Arm/Group | Phase 2 Arm A1: TCZ +/- nbDMARD Once Per Week (qw) | Phase 2 Arm A2: TCZ +/- nbDMARD Every Two Weeks (q2w)
Number analyzed (Participants) | 89 | 90
SJC
  Baseline values | 9.28 (6.52) | 9.23 (7.55)
  Week 28: number analyzed (Participants) | 88 | 90
  Week 28 | -8.64 (6.19) | -8.14 (6.81)
  Week 32: number analyzed (Participants) | 87 | 90
  Week 32 | -8.54 (7.02) | -8.62 (7.13)
  Week 36: number analyzed (Participants) | 86 | 89
  Week 36 | -8.48 (6.50) | -8.38 (6.76)
  Week 40: number analyzed (Participants) | 84 | 88
  Week 40 | -8.85 (6.40) | -8.51 (6.59)
  Week 44: number analyzed (Participants) | 82 | 89
  Week 44 | -8.73 (6.62) | -8.62 (6.97)
  Week 48: number analyzed (Participants) | 84 | 89
  Week 48 | -9.06 (6.58) | -8.72 (7.34)
  LOCF visit | -8.82 (6.51) | -8.64 (7.33)

17. Secondary Outcome: Percentages of Patients Who Achieve DAS28-ESR Remission (DAS28 < 2.6) up to Week 48
Description: as for outcome 1
Time Frame: Week 48
Population: Analysis was conducted on the FAS
Measure: Mean (95% Confidence Interval); unit: Percentage of participants
Groups:
- Phase 2 Arm A1 - Monotherapy - qw: Participants who achieved sustained clinical remission (DAS28-ESR <2.6) at Week 20 and Week 24 in Part 1 were randomized to tocilizumab given every week monotherapy from Week 24 to Week 48.
- Phase 2 Arm A1- Combination Therapy - qw: Participants who achieved sustained clinical remission (DAS28-ESR <2.6) at Week 20 and Week 24 in Part 1 were randomized to tocilizumab given every week in combination with methotrexate or other non-biologics DMARDs from Week 24 to Week 48.
- Phase 2 Arm A2 - Monotherapy - q2w: Participants who achieved sustained clinical remission (DAS28-ESR <2.6) at Week 20 and Week 24 in Part 1 were randomized to tocilizumab given every 2 weeks monotherapy from Week 24 to Week 48.
- Phase 2 Arm A2 - Combination Therapy - q2w: Participants who achieved sustained clinical remission (DAS28-ESR <2.6) at Week 20 and Week 24 in Part 1 were randomized to tocilizumab given every 2 weeks in combination with methotrexate or other non-biologics DMARDs from Week 24 to Week 48.
Arm/Group | Phase 2 Arm A1 - Monotherapy - qw | Phase 2 Arm A1- Combination Therapy - qw | Phase 2 Arm A2 - Monotherapy - q2w | Phase 2 Arm A2 - Combination Therapy - q2w
Number analyzed (Participants) | 23 | 66 | 23 | 67
Percentage of participants
  Week 28: number analyzed (Participants) | 23 | 65 | 23 | 67
  Week 28 | 82.6 [61.22 to 95.05] | 90.6 [80.70 to 96.48] | 87.0 [66.41 to 97.22] | 83.1 [71.73 to 91.24]
  Week 32: number analyzed (Participants) | 22 | 65 | 23 | 67
  Week 32 | 81.8 [59.72 to 94.81] | 89.1 [78.75 to 95.49] | 78.3 [56.30 to 92.54] | 82.1 [70.80 to 90.39]
  Week 36: number analyzed (Participants) | 21 | 65 | 23 | 67
  Week 36 | 90.5 [69.62 to 98.83] | 76.9 [64.81 to 86.47] | 86.4 [65.09 to 97.09] | 86.4 [75.69 to 93.57]
  Week 40: number analyzed (Participants) | 20 | 64 | 23 | 67
  Week 40 | 85.0 [62.11 to 96.79] | 81.3 [69.54 to 89.92] | 77.3 [54.63 to 92.18] | 81.8 [70.39 to 90.24]
  Week 44: number analyzed (Participants) | 19 | 63 | 23 | 67
  Week 44 | 94.7 [73.97 to 99.87] | 87.3 [76.50 to 94.35] | 77.3 [54.63 to 92.18] | 78.8 [66.98 to 87.89]
  Week 48: number analyzed (Participants) | 20 | 64 | 23 | 67
  Week 48 | 100 [NA to NA] — CI unavailable because the central value is 100% | 89.1 [78.75 to 95.49] | 77.3 [54.63 to 92.18] | 72.7 [60.36 to 82.97]
  LOCF Visit | 91.3 [71.96 to 98.93] | 89.4 [79.36 to 95.63] | 73.9 [51.59 to 89.77] | 73.1 [60.90 to 83.24]

18. Secondary Outcome: Percentages of Patients With Remission (CDAI<2.8) Until Week 24
Description: as for outcome 9
Time Frame: From baseline to Week 24
Population: Analysis was conducted on the FAS
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Phase 1: Tocilizumab Monotherapy | Phase 1: Combination Therapy
Number analyzed (Participants) | 74 | 327
Percentage of participants
  Baseline visit | 0 [0 to 0] | 0 [0 to 0]
  Week 2: number analyzed (Participants) | 74 | 319
  Week 2 | 2.7 [0.33 to 9.42] | 1.6 [0.51 to 3.62]
  Week 4: number analyzed (Participants) | 73 | 312
  Week 4 | 2.7 [0.33 to 9.55] | 5.1 [2.96 to 8.19]
  Week 8: number analyzed (Participants) | 73 | 300
  Week 8 | 11.0 [4.85 to 20.46] | 14.4 [10.61 to 18.88]
  Week 12: number analyzed (Participants) | 70 | 296
  Week 12 | 15.7 [8.11 to 26.38] | 19.3 [14.92 to 24.22]
  Week 16: number analyzed (Participants) | 69 | 292
  Week 16 | 18.8 [10.43 to 30.06] | 22.8 [18.06 to 28.02]
  Week 20: number analyzed (Participants) | 65 | 284
  Week 20 | 27.7 [17.31 to 40.19] | 26.8 [21.70 to 32.31]
  Week 24: number analyzed (Participants) | 64 | 281
  Week 24 | 29.7 [18.91 to 42.42] | 30.2 [24.93 to 35.99]
  LOCF visit | 29.7 [19.66 to 41.48] | 29.4 [24.48 to 34.62]

19. Secondary Outcome: Percentages of Patients With Remission (CDAI<2.8) Until Week 48
Description: as for outcome 9
Time Frame: From week 28 until week 48
Population: Analysis was conducted on the FAS
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Phase 2 Arm A1: TCZ +/- nbDMARD Once Per Week (qw) | Phase 2 Arm A2: TCZ +/- nbDMARD Every Two Weeks (q2w)
Number analyzed (Participants) | 89 | 90
Percentage of participants
  Week 28: number analyzed (Participants) | 88 | 90
  Week 28 | 46.6 [35.88 to 57.54] | 48.3 [37.59 to 59.16]
  Week 32: number analyzed (Participants) | 87 | 90
  Week 32 | 48.3 [37.42 to 59.25] | 45.6 [35.02 to 56.40]
  Week 36: number analyzed (Participants) | 86 | 89
  Week 36 | 52.3 [41.27 to 63.21] | 46.6 [35.88 to 57.54]
  Week 40: number analyzed (Participants) | 84 | 88
  Week 40 | 52.4 [41.19 to 63.40] | 45.5 [34.80 to 56.42]
  Week 44: number analyzed (Participants) | 82 | 89
  Week 44 | 50.0 [38.75 to 61.25] | 50.6 [39.75 to 61.33]
  Week 48: number analyzed (Participants) | 84 | 89
  Week 48 | 59.0 [47.69 to 69.72] | 53.9 [43.04 to 64.56]
  LOCF Visit | 57.8 [46.91 to 68.12] | 60.3 [52.77 to 67.56]

20. Secondary Outcome: Percentages of Patients With Remission (SDAI<3.3) Until Week 24
Description: as for outcome 11
Time Frame: From baseline to Week 24
Population: Analysis was conducted on the FAS
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Phase 1: Tocilizumab Monotherapy | Phase 1: Combination Therapy
Number analyzed (Participants) | 74 | 327
Percentage of participants
  Baseline visit | 0 [0 to 0] | 0 [0 to 0]
  Week 2: number analyzed (Participants) | 74 | 319
  Week 2 | 1.4 [0.04 to 7.50] | 1.9 [0.71 to 4.14]
  Week 4: number analyzed (Participants) | 73 | 312
  Week 4 | 2.9 [0.35 to 9.94] | 4.8 [2.72 to 7.83]
  Week 8: number analyzed (Participants) | 73 | 300
  Week 8 | 11.1 [4.92 to 20.72] | 14.6 [10.75 to 19.13]
  Week 12: number analyzed (Participants) | 70 | 296
  Week 12 | 14.3 [7.07 to 24.71] | 18.8 [14.47 to 23.72]
  Week 16: number analyzed (Participants) | 69 | 292
  Week 16 | 17.4 [9.32 to 28.41] | 22.2 [17.56 to 27.47]
  Week 20: number analyzed (Participants) | 65 | 284
  Week 20 | 28.1 [17.60 to 40.76] | 25.8 [20.77 to 31.36]
  Week 24: number analyzed (Participants) | 64 | 281
  Week 24 | 31.7 [20.58 to 44.69] | 28.8 [23.53 to 34.49]
  LOCF visit | 28.4 [18.50 to 40.05] | 25.4 [20.75 to 30.46]

21. Secondary Outcome: Percentages of Patients With Remission (SDAI<3.3) Until Week 48
Description: as for outcome 11
Time Frame: From week 28 until week 48
Population: Analysis was conducted on the FAS
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Phase 2 Arm A1: TCZ +/- nbDMARD Once Per Week (qw) | Phase 2 Arm A2: TCZ +/- nbDMARD Every Two Weeks (q2w)
Number analyzed (Participants) | 89 | 90
Percentage of participants
  Week 28: number analyzed (Participants) | 88 | 90
  Week 28 | 50.0 [39.02 to 60.98] | 46.0 [35.23 to 57.00]
  Week 32: number analyzed (Participants) | 87 | 90
  Week 32 | 48.8 [37.90 to 59.86] | 45.6 [35.02 to 56.40]
  Week 36: number analyzed (Participants) | 86 | 89
  Week 36 | 53.5 [42.41 to 64.32] | 47.7 [36.96 to 58.65]
  Week 40: number analyzed (Participants) | 84 | 88
  Week 40 | 55.4 [44.10 to 66.34] | 44.3 [33.73 to 55.30]
  Week 44: number analyzed (Participants) | 82 | 89
  Week 44 | 50.0 [38.75 to 61.25] | 47.2 [36.51 to 58.06]
  Week 48: number analyzed (Participants) | 84 | 89
  Week 48 | 52.4 [41.11 to 63.59] | 47.7 [36.96 to 58.65]
  LOCF Visit | 51.7 [40.48 to 62.41] | 47.8 [37.13 to 58.57]

22. Secondary Outcome: Percentage of Patients Who Achieve Low Disease Activity Based on DAS28-ESR Criteria (DAS28-ESR </=3.2) up to Week 24
Description: The DAS28 is a combined index for measuring disease activity in RA. The index includes the assessment of 28 joints for swelling and tenderness, acute phase response (ESR or CRP), and general health status. For this study ESR is used to calculate the DAS28 score.
Time Frame: From baseline to Week 24
Population: Analysis was conducted on the FAS.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Phase 1: Tocilizumab Monotherapy | Phase 1: Combination Therapy
Number analyzed (Participants) | 74 | 327
Percentage of participants
  Week 2: number analyzed (Participants) | 74 | 319
  Week 2 | 21.6 [12.89 to 32.72] | 21.5 [17.12 to 26.47]
  Week 4: number analyzed (Participants) | 73 | 300
  Week 4 | 26.0 [16.45 to 37.62] | 36.8 [31.39 to 42.41]
  Week 8 | 50.7 [38.72 to 62.60] | 55.4 [49.54 to 61.16]
  Week 12: number analyzed (Participants) | 70 | 296
  Week 12 | 58.6 [46.17 to 70.23] | 67.7 [62.01 to 73.00]
  Week 16: number analyzed (Participants) | 69 | 292
  Week 16 | 66.7 [54.29 to 77.56] | 72.4 [66.89 to 77.48]
  Week 20: number analyzed (Participants) | 65 | 284
  Week 20 | 67.7 [54.95 to 78.77] | 78.2 [72.91 to 82.83]
  Week 24: number analyzed (Participants) | 64 | 281
  Week 24 | 75.0 [62.60 to 84.98] | 81.1 [75.98 to 85.49]
  LOCF visit | 73.0 [61.39 to 82.65] | 74.0 [68.90 to 78.68]

23. Secondary Outcome: Percentage of Patients Who Achieve Low Disease Activity Based on DAS28-ESR Criteria (DAS28-ESR </=3.2) up to Week 48
Description: The DAS28 is a combined index for measuring disease activity in RA. The index includes the assessment of 28 joints for swelling and tenderness, acute phase response (ESR or CRP), and general health status. For this study ESR was used to calculate the DAS28 score.
Time Frame: From week 28 until week 48
Population: Analysis was conducted on the FAS.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Phase 2 Arm A1: TCZ +/- nbDMARD Once Per Week (qw) | Phase 2 Arm A2: TCZ +/- nbDMARD Every Two Weeks (q2w)
Number analyzed (Participants) | 89 | 90
Percentage of participants
  Week 28: number analyzed (Participants) | 88 | 90
  Week 28 | 95.4 [88.64 to 98.73] | 88.6 [80.09 to 94.41]
  Week 32: number analyzed (Participants) | 87 | 90
  Week 32 | 91.9 [83.95 to 96.66] | 92.2 [84.63 to 96.82]
  Week 36: number analyzed (Participants) | 86 | 89
  Week 36 | 87.2 [78.27 to 93.44] | 92.0 [84.30 to 96.74]
  Week 40: number analyzed (Participants) | 84 | 88
  Week 40 | 89.3 [80.63 to 94.98] | 92.0 [84.30 to 96.74]
  Week 44: number analyzed (Participants) | 82 | 89
  Week 44 | 96.3 [89.68 to 99.24] | 87.5 [78.73 to 93.59]
  Week 48: number analyzed (Participants) | 84 | 89
  Week 48 | 95.1 [87.98 to 98.66] | 86.4 [77.39 to 92.75]
  LOCF Visit | 94.4 [87.37 to 98.15] | 85.6 [76.57 to 92.08]

24. Secondary Outcome: Percentage of Patients Who Achieve Low Disease Activity Based on CDAI Score (CDAI<10) Until Week 24
Description: as for outcome 9
Time Frame: From baseline to Week 24
Population: Analysis was conducted on the FAS.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Phase 1: Tocilizumab Monotherapy | Phase 1: Combination Therapy
Number analyzed (Participants) | 74 | 327
Percentage of participants
  Week 2: number analyzed (Participants) | 74 | 319
  Week 2 | 13.5 [6.68 to 23.45] | 16.9 [12.98 to 21.50]
  Week 4: number analyzed (Participants) | 73 | 312
  Week 4 | 24.7 [15.32 to 36.14] | 26.9 [22.08 to 32.21]
  Week 8: number analyzed (Participants) | 73 | 300
  Week 8 | 41.1 [29.71 to 53.23] | 47.5 [41.71 to 53.32]
  Week 12: number analyzed (Participants) | 70 | 296
  Week 12 | 57.1 [44.75 to 68.91] | 52.4 [46.51 to 58.17]
  Week 16: number analyzed (Participants) | 69 | 292
  Week 16 | 62.3 [49.83 to 73.71] | 60.7 [54.81 to 66.35]
  Week 20: number analyzed (Participants) | 65 | 284
  Week 20 | 66.2 [53.35 to 77.43] | 65.1 [59.29 to 70.68]
  Week 24: number analyzed (Participants) | 64 | 281
  Week 24 | 71.9 [59.24 to 82.40] | 66.9 [61.07 to 72.38]
  LOCF visit | 66.2 [54.28 to 76.81] | 61.2 [55.64 to 66.48]

25. Secondary Outcome: Percentage of Patients Who Achieve Low Disease Activity Based on CDAI Score (CDAI<10) Until Week 48
Description: as for outcome 9
Time Frame: From week 28 until week 48
Population: Analysis was conducted on the FAS.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Phase 2 Arm A1: TCZ +/- nbDMARD Once Per Week (qw) | Phase 2 Arm A2: TCZ +/- nbDMARD Every Two Weeks (q2w)
Number analyzed (Participants) | 89 | 90
Percentage of participants
  Week 28: number analyzed (Participants) | 88 | 90
  Week 28 | 86.4 [77.39 to 92.75] | 85.4 [76.32 to 91.99]
  Week 32: number analyzed (Participants) | 87 | 90
  Week 32 | 89.7 [81.27 to 95.16] | 86.7 [77.87 to 92.92]
  Week 36: number analyzed (Participants) | 86 | 89
  Week 36 | 80.2 [70.25 to 88.04] | 89.8 [81.47 to 95.22]
  Week 40: number analyzed (Participants) | 84 | 88
  Week 40 | 86.9 [77.78 to 93.28] | 88.6 [80.09 to 94.41]
  Week 44: number analyzed (Participants) | 82 | 89
  Week 44 | 89.0 [80.18 to 94.86] | 85.4 [76.32 to 91.99]
  Week 48: number analyzed (Participants) | 84 | 89
  Week 48 | 92.8 [84.93 to 97.30] | 87.6 [78.96 to 93.67]
  LOCF Visit | 91.0 [83.05 to 96.04] | 87.8 [79.18 to 93.74]

26. Secondary Outcome: Percentage of Patients Who Achieved Low Disease Activity (LDA) Based on SDAI Score (SDAI<11) Until Week 24
Description: as for outcome 11
Time Frame: From baseline to Week 24
Population: Analysis was conducted on the FAS.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Phase 1: Tocilizumab Monotherapy | Phase 1: Combination Therapy
Number analyzed (Participants) | 74 | 327
Percentage of participants
  Week 2: number analyzed (Participants) | 74 | 319
  Week 2 | 16.7 [8.92 to 27.30] | 17.6 [13.56 to 22.32]
  Week 4: number analyzed (Participants) | 73 | 312
  Week 4 | 27.1 [17.20 to 39.10] | 28.3 [23.36 to 33.65]
  Week 8: number analyzed (Participants) | 73 | 300
  Week 8 | 41.7 [30.15 to 53.89] | 48.1 [42.31 to 54.00]
  Week 12: number analyzed (Participants) | 70 | 296
  Week 12 | 58.6 [46.17 to 70.23] | 55.6 [49.74 to 61.41]
  Week 16: number analyzed (Participants) | 69 | 292
  Week 16 | 63.8 [51.31 to 75.01] | 62.5 [56.63 to 68.11]
  Week 20: number analyzed (Participants) | 65 | 284
  Week 20 | 65.6 [52.70 to 77.05] | 66.3 [60.43 to 71.83]
  Week 24: number analyzed (Participants) | 64 | 281
  Week 24 | 74.6 [62.06 to 84.73] | 67.3 [61.41 to 72.75]
  LOCF visit | 63.5 [51.51 to 74.40] | 56.9 [51.32 to 62.32]

27. Secondary Outcome: Percentage of Patients Who Achieved Low Disease Activity (LDA) Based on SDAI Score (SDAI<11) Until Week 48
Description: as for outcome 11
Time Frame: From week 28 until week 48
Population: Analysis was conducted on the FAS.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Phase 2 Arm A1: TCZ +/- nbDMARD Once Per Week (qw) | Phase 2 Arm A2: TCZ +/- nbDMARD Every Two Weeks (q2w)
Number analyzed (Participants) | 89 | 90
Percentage of participants
  Week 28: number analyzed (Participants) | 88 | 90
  Week 28 | 84.9 [75.54 to 91.70] | 83.89 [74.48 to 90.91]
  Week 32: number analyzed (Participants) | 87 | 90
  Week 32 | 89.5 [81.06 to 95.10] | 85.6 [76.57 to 92.08]
  Week 36: number analyzed (Participants) | 86 | 89
  Week 36 | 79.1 [68.95 to 87.10] | 87.5 [78.73 to 93.59]
  Week 40: number analyzed (Participants) | 84 | 88
  Week 40 | 86.7 [77.52 to 93.19] | 86.4 [77.39 to 92.75]
  Week 44: number analyzed (Participants) | 82 | 89
  Week 44 | 91.5 [83.20 to 96.50] | 82.0 [72.45 to 89.36]
  Week 48: number analyzed (Participants) | 84 | 89
  Week 48 | 93.9 [86.34 to 97.99] | 81.8 [72.16 to 89.24]
  LOCF Visit | 91.0 [83.05 to 96.04] | 81.1 [71.49 to 88.59]

28. Secondary Outcome: Safety: Number of Patients Reporting Adverse Events up to Week 24
Description: Number of patients reporting any treatment emergent adverse event (TEAE), at least one TEAE of special interest, at least one serious TEAE, at least one TEAE leading to dose modification, at least one TEAE leading to discontinuation up to week 24
Time Frame: From baseline to Week 24
Population: Analysis was conducted on the FAS.
Measure: Number; unit: Number of participants
Arm/Group | Phase 1: Tocilizumab Monotherapy | Phase 1: Combination Therapy
Number analyzed (Participants) | 74 | 327
Number of participants
  Any treatment emergent adverse event (TEAE) | 52 | 254
  At least one TEAE of special interest | 2 | 13
  At least one serious TEAE | 3 | 10
  At least one TEAE leading to dose modification | 24 | 103
  At least one TEAE leading to discontinuation | 4 | 21

29. Secondary Outcome: Safety: Number of Patients Reporting Adverse Events up to Week 48
Description: Number of patients reporting any treatment emergent adverse event (TEAE), at least one TEAE of special interest, at least one serious TEAE, at least one TEAE leading to dose modification, at least one TEAE leading to discontinuation up to week 48
Time Frame: From week 24 until week 48
Population: Analysis was conducted on the FAS.
Measure: Number; unit: Number of participants
Groups:
- Phase 2 Arm D: Non Responders: Patients who didn't achieve any therapeutic response up to week 24 and were discontinued from the study.
Arm/Group | Phase 2 Arm A1: TCZ +/- nbDMARD Once Per Week (qw) | Phase 2 Arm A2: TCZ +/- nbDMARD Every Two Weeks (q2w) | Phase 2 Arm B: Participants With Low Disease Activity | Phase 2 Arm C: Moderate EULAR Response at Week 24 | Phase 2 Arm D: Non Responders
Number analyzed (Participants) | 89 | 90 | 95 | 67 | 2
Number of participants
  Any TEAE | 50 | 63 | 68 | 46 | 1
  At least one TEAE of special interest | 1 | 2 | 2 | 4 | 0
  At least one serious TEAE | 2 | 1 | 2 | 5 | 1
  At least one TEAE leading to dose modification | 15 | 23 | 23 | 21 | 1
  At least one TEAE leading to discontinuation | 0 | 0 | 0 | 2 | 0

30. Secondary Outcome: Immunogenicity: Number of Patients With Anti-tocilizumab Antibodies up to Week 24
Description: Number of patients resulting positive to anti-tocilizumab antibodies test are reported.
Time Frame: From baseline to Week 24
Population: Analysis was conducted on the FAS.
Measure: Number; unit: Number of participants
Arm/Group | Phase 1: Tocilizumab Monotherapy | Phase 1: Combination Therapy
Number analyzed (Participants) | 74 | 327
Number of participants
  Screen - Baseline | 6 | 13
  Screen - Week 12 | 1 | 2
  Screen - Week 24 | 3 | 9
  Confirmatory - Baseline | 4 | 5
  Confirmatory - Week 12 | 1 | 0
  Confirmatory - Week 24 | 1 | 3

31. Secondary Outcome: Immunogenicity: Number of Patients With Anti-tocilizumab Antibodies up to Week 48
Description: Number of patients resulting positive to anti-tocilizumab antibodies test are reported.
Time Frame: From week 24 until week 48
Population: Analysis was conducted on the FAS.
Measure: Number; unit: Number of participants
Arm/Group | Phase 2 Arm A1: TCZ +/- nbDMARD Once Per Week (qw) | Phase 2 Arm A2: TCZ +/- nbDMARD Every Two Weeks (q2w) | Phase 2 Arm B: Participants With Low Disease Activity | Phase 2 Arm C: Moderate EULAR Response at Week 24 | Phase 2 Arm D: Non Responders
Number analyzed (Participants) | 89 | 90 | 95 | 67 | 2
Number of participants
  Screen - Week 36: number analyzed (Participants) | 86 | 89 | 91 | 59 | 0
  Screen - Week 36 | 0 | 0 | 0 | 2 |
  Screen - Week 48: number analyzed (Participants) | 84 | 89 | 89 | 59 | 0
  Screen - Week 48 | 1 | 3 | 2 | 3 |
  Confirmatory - Week 36: number analyzed (Participants) | 86 | 89 | 88 | 59 | 0
  Confirmatory - Week 36 | 0 | 0 | 0 | 1 |
  Confirmatory - Week 48: number analyzed (Participants) | 84 | 89 | 88 | 59 | 0
  Confirmatory - Week 48 | 0 | 0 | 0 | 1 |

32. Secondary Outcome: Immunogenicity: TCZ Levels up to Week 24
Description: Mean concentrations of TCZ in patients' blood are reported.
Time Frame: From baseline to Week 24
Population: Analysis was conducted on the FAS.
Measure: Mean (Standard Deviation); unit: mcg/ml
Arm/Group | Phase 1: Tocilizumab Monotherapy | Phase 1: Combination Therapy
Number analyzed (Participants) | 74 | 327
mcg/ml
  Baseline: number analyzed (Participants) | 1 | 4
  Baseline | 0.49 (NA) — Analysis was done for one participant only. | 0.67 (0.34)
  Week 12: number analyzed (Participants) | 67 | 285
  Week 12 | 37.97 (20.11) | 41.23 (20.89)
  Week 24: number analyzed (Participants) | 62 | 273
  Week 24 | 46.42 (28.35) | 46.87 (27.65)

33. Secondary Outcome: Immunogenicity: TCZ Levels at Week 36 and Early Withdrawal Visit
Description: Mean concentrations of TCZ in patients' blood are reported.
Time Frame: week 36 and early withdrawal visit
Population: Analysis was conducted on the FAS.
Measure: Mean (Standard Deviation); unit: mcg/ml
Groups:
- Phase 2 Arm B: Participants With Low Disease Activity: Participants who did not achieve sustained clinical remission at Week 20 and Week 24 but achieve low disease activity (DAS 28-ESR ≤ 3.2) at Week 24 continued with initial treatment of tocilizumab as a single fixed dose monotherapy or in combination with methotrexate or other non-biologics DMARDs from Week 24 to Week 48. Participants who achieved moderate EULAR response at Week 24 continued in the study with initial treatment as per investigator's judgement.
Arm/Group | Phase 2 Arm A1: TCZ +/- nbDMARD Once Per Week (qw) | Phase 2 Arm A2: TCZ +/- nbDMARD Every Two Weeks (q2w) | Phase 2 Arm B: Participants With Low Disease Activity | Phase 2 Arm C: Moderate EULAR Response at Week 24 | Phase 2 Arm D: Non Responders
Number analyzed (Participants) | 89 | 90 | 95 | 67 | 2
mcg/ml
  Week 36: number analyzed (Participants) | 84 | 86 | 86 | 55 | 0
  Week 36 | 48.47 (30.17) | 16.77 (16.10) | 41.89 (28.82) | 48.33 (25.79) |
  Early withdrawal visit: number analyzed (Participants) | 2 | 1 | 4 | 2 | 1
  Early withdrawal visit | 36.45 (18.03) | 19.20 (NA) — Analysis was conducted for one participant only | 24.43 (20.83) | 13.75 (4.60) | 1.78 (NA) — Analysis was conducted for one participant only

34. Secondary Outcome: Immunogenicity: SIL-6R Levels up to Week 24
Description: Mean concentration of SIL-6R in patients' blood are reported.
Time Frame: From baseline to Week 24
Population: Analysis was conducted on the FAS.
Measure: Mean (Standard Deviation); unit: mcg/ml
Arm/Group | Phase 1: Tocilizumab Monotherapy | Phase 1: Combination Therapy
Number analyzed (Participants) | 74 | 327
mcg/ml
  Baseline: number analyzed (Participants) | 74 | 321
  Baseline | 42.85 (16.26) | 39.29 (11.10)
  Week 12: number analyzed (Participants) | 69 | 290
  Week 12 | 566.47 (210.49) | 570.34 (228.54)
  Week 24: number analyzed (Participants) | 63 | 279
  Week 24 | 570.49 (198.26) | 565.34 (198.32)

35. Secondary Outcome: Immunogenicity: SIL-6R Levels at Week 36 and Early Withdrawal Visit
Description: Mean concentration of SIL-6R in patients' blood are reported.
Time Frame: Baseline, Week 36 and Early Withdrawal Visit
Population: Analysis was conducted on the FAS.
Measure: Mean (Standard Deviation); unit: mcg/ml
Arm/Group | Phase 2 Arm A1: TCZ +/- nbDMARD Once Per Week (qw) | Phase 2 Arm A2: TCZ +/- nbDMARD Every Two Weeks (q2w) | Phase 2 Arm B: Participants With Low Disease Activity | Phase 2 Arm C: Moderate EULAR Response at Week 24 | Phase 2 Arm D: Non Responders
Number analyzed (Participants) | 89 | 90 | 95 | 67 | 2
mcg/ml
  Baseline: number analyzed (Participants) | 88 | 88 | 94 | 67 | 2
  Baseline | 39.87 (10.46) | 39.70 (16.46) | 39.39 (11.24) | 43.11 (11.85) | 37.30 (11.46)
  Week 36: number analyzed (Participants) | 86 | 89 | 88 | 59 | 0
  Week 36 | 539.89 (152.71) | 476.28 (156.50) | 542.99 (168.30) | 552.65 (184.21) |
  Early withdrawal visit: number analyzed (Participants) | 3 | 1 | 6 | 5 | 1
  Early withdrawal visit | 412.53 (323.49) | 643.00 (NA) — Analysis was conducted on one participant only. | 338.38 (230.82) | 217.74 (236.21) | 513.00 (NA) — Analysis was conducted on one participant only.

36. Secondary Outcome: Patient Global Assessment of Disease Activity Visual Analogue Scale (VAS) up to Week 24
Description: This patient reported outcome assessment represents the patient's overall assessment of their current disease activity on a 100 mm horizontal VAS. The extreme left end of the line should be described as "no disease activity" (symptom-free and no arthritis symptoms) and the extreme right end as "maximum disease activity" (maximum arthritis disease activity). The line was marked by the participant and the distance from the left edge was recorded and the mean values are reported.
Time Frame: From baseline to Week 24
Population: Analysis was conducted on the FAS.
Measure: Mean (Standard Deviation); unit: Millimeters
Arm/Group | Phase 1: Tocilizumab Monotherapy | Phase 1: Combination Therapy
Number analyzed (Participants) | 74 | 327
Millimeters
  Baseline: number analyzed (Participants) | 74 | 319
  Baseline | 65.26 (19.77) | 59.40 (17.61)
  Week 2: number analyzed (Participants) | 74 | 319
  Week 2 | 49.53 (22.78) | 44.16 (21.97)
  Week 4: number analyzed (Participants) | 73 | 312
  Week 4 | 38.21 (22.92) | 35.19 (20.83)
  Week 8: number analyzed (Participants) | 73 | 300
  Week 8 | 30.03 (21.65) | 26.04 (20.59)
  Week 12: number analyzed (Participants) | 70 | 296
  Week 12 | 22.71 (18.56) | 22.24 (17.97)
  Week 16: number analyzed (Participants) | 69 | 291
  Week 16 | 19.28 (18.22) | 20.71 (18.65)
  Week 20: number analyzed (Participants) | 65 | 284
  Week 20 | 16.80 (16.68) | 18.79 (17.79)
  Week 24: number analyzed (Participants) | 64 | 281
  Week 24 | 16.63 (15.19) | 19.00 (18.36)
  LOCF visit | 20.36 (19.25) | 22.23 (20.86)

37. Secondary Outcome: Patient Global Assessment of Disease Activity Visual Analogue Scale (VAS) up to Week 48
Description: as for outcome 36
Time Frame: Baseline, from week 28 until week 48
Population: Analysis was conducted on the FAS.
Measure: Mean (Standard Deviation); unit: Millimeters
Arm/Group | Phase 2 Arm A1: TCZ +/- nbDMARD Once Per Week (qw) | Phase 2 Arm A2: TCZ +/- nbDMARD Every Two Weeks (q2w)
Number analyzed (Participants) | 89 | 90
Millimeters
  Baseline | 58.97 (17.40) | 60.96 (20.13)
  Week 28: number analyzed (Participants) | 88 | 90
  Week 28 | 11.97 (14.10) | 12.74 (15.07)
  Week 32: number analyzed (Participants) | 87 | 90
  Week 32 | 10.78 (15.33) | 10.80 (11.36)
  Week 36: number analyzed (Participants) | 86 | 89
  Week 36 | 11.99 (16.23) | 10.30 (13.20)
  Week 40: number analyzed (Participants) | 84 | 88
  Week 40 | 10.62 (13.49) | 10.94 (14.12)
  Week 44: number analyzed (Participants) | 82 | 89
  Week 44 | 9.50 (11.30) | 10.06 (12.14)
  Week 48: number analyzed (Participants) | 84 | 89
  Week 48 | 8.13 (10.52) | 9.99 (13.88)
  LOCF visit | 8.97 (11.63) | 10.21 (13.96)

38. Secondary Outcome: Assessment of Pain Reported by the Patient (VAS) Until Week 24
Description: This patient reported outcome assessment represents the patient's assessment of his/her current level of pain on a 100 mm horizontal VAS. The extreme left end of the line should be described as "no pain" and the extreme right end as "unbearable pain".
Time Frame: From baseline to Week 24
Population: Analysis was conducted on the FAS.
Measure: Mean (Standard Deviation); unit: Millimeters
Arm/Group | Phase 1: Tocilizumab Monotherapy | Phase 1: Combination Therapy
Number analyzed (Participants) | 74 | 327
Millimeters
  Baseline | 66.38 (20.70) | 58.59 (23.70)
  Week 2: number analyzed (Participants) | 74 | 319
  Week 2 | 53.20 (24.43) | 47.46 (25.14)
  Week 4: number analyzed (Participants) | 73 | 312
  Week 4 | 43.11 (24.69) | 42.88 (24.57)
  Week 8: number analyzed (Participants) | 73 | 300
  Week 8 | 35.95 (24.62) | 34.28 (25.94)
  Week 12: number analyzed (Participants) | 70 | 296
  Week 12 | 29.44 (22.37) | 31.07 (24.97)
  Week 16: number analyzed (Participants) | 69 | 292
  Week 16 | 32.17 (22.01) | 30.18 (24.00)
  Week 20: number analyzed (Participants) | 65 | 284
  Week 20 | 26.58 (22.13) | 28.26 (24.16)
  Week 24: number analyzed (Participants) | 64 | 281
  Week 24 | 23.56 (21.17) | 26.43 (23.30)
  LOCF visit | 27.34 (24.41) | 29.78 (25.18)

39. Secondary Outcome: Assessment of Pain Reported by the Patient (VAS) Until Week 48
Description: as for outcome 38
Time Frame: Baseline, from week 28 until week 48
Population: Analysis was conducted on the FAS.
Measure: Mean (Standard Deviation); unit: Millimeters
Arm/Group | Phase 2 Arm A1: TCZ +/- nbDMARD Once Per Week (qw) | Phase 2 Arm A2: TCZ +/- nbDMARD Every Two Weeks (q2w)
Number analyzed (Participants) | 89 | 90
Millimeters
  Baseline | 55.73 (21.68) | 56.00 (23.56)
  Week 28: number analyzed (Participants) | 88 | 90
  Week 28 | 17.33 (20.14) | 15.67 (17.65)
  Week 32: number analyzed (Participants) | 87 | 90
  Week 32 | 17.08 (20.47) | 17.27 (17.69)
  Week 36: number analyzed (Participants) | 86 | 88
  Week 36 | 18.81 (23.88) | 14.36 (15.65)
  Week 40: number analyzed (Participants) | 84 | 88
  Week 40 | 16.96 (20.89) | 17.07 (17.86)
  Week 44: number analyzed (Participants) | 82 | 89
  Week 44 | 15.05 (18.02) | 16.27 (17.70)
  Week 48: number analyzed (Participants) | 84 | 89
  Week 48 | 11.90 (15.56) | 16.31 (19.85)
  LOCF visit | 12.74 (15.99) | 16.41 (19.76)

40. Secondary Outcome: Health Assessment Questionnaire-Disability Index (HAQ-DI) up to Week 24
Description: The Stanford HAQ-DI is a patient-oriented outcome assessment questionnaire specific for RA. It consists of 20 questions referring to eight component sets: dressing/grooming, arising, eating, walking, hygiene, reach, grip, and activities.
  To respond to each question, a four-level response (score of 0 to 3 points), with higher scores showing larger functional limitations, was chosen. Scoring was as follows with respect to performance of participant's everyday activities: 0 (equals)=without difficulties; 1=with some difficulties; 2=with great difficulties; and 3=unable to perform these actions at all. Minimum score was 0, maximum score was 3.
Time Frame: From baseline to Week 24
Population: Analysis was conducted on the FAS.
Measure: Mean (Standard Deviation); unit: HAQ-DI score
Arm/Group | Phase 1: Tocilizumab Monotherapy | Phase 1: Combination Therapy
Number analyzed (Participants) | 74 | 327
HAQ-DI score
  Baseline: number analyzed (Participants) | 74 | 324
  Baseline | 1.49 (0.76) | 1.36 (0.70)
  Week 2: number analyzed (Participants) | 73 | 317
  Week 2 | 1.39 (0.74) | 1.18 (0.69)
  Week 4: number analyzed (Participants) | 72 | 309
  Week 4 | 1.20 (0.74) | 1.05 (0.69)
  Week 8: number analyzed (Participants) | 73 | 300
  Week 8 | 1.10 (0.75) | 0.95 (0.71)
  Week 12: number analyzed (Participants) | 69 | 295
  Week 12 | 0.99 (0.74) | 0.91 (0.71)
  Week 16: number analyzed (Participants) | 69 | 292
  Week 16 | 0.99 (0.72) | 0.87 (0.70)
  Week 20: number analyzed (Participants) | 65 | 283
  Week 20 | 0.88 (0.70) | 0.83 (0.71)
  Week 24: number analyzed (Participants) | 63 | 281
  Week 24 | 0.85 (0.71) | 0.82 (0.70)
  LOCF visit | 0.97 (0.76) | 0.88 (0.73)

41. Secondary Outcome: Health Assessment Questionnaire-Disability Index (HAQ-DI) up to Week 48
Description: as for outcome 40
Time Frame: Baseline, from week 28 until week 48
Population: Analysis was conducted on the FAS.
Measure: Mean (Standard Deviation); unit: HAQ-DI score
Arm/Group | Phase 2 Arm A1: TCZ +/- nbDMARD Once Per Week (qw) | Phase 2 Arm A2: TCZ +/- nbDMARD Every Two Weeks (q2w)
Number analyzed (Participants) | 89 | 90
HAQ-DI score
  Baseline: number analyzed (Participants) | 88 | 89
  Baseline | 1.21 (0.68) | 1.20 (0.70)
  Week 28: number analyzed (Participants) | 88 | 90
  Week 28 | 0.58 (0.56) | 0.57 (0.64)
  Week 32: number analyzed (Participants) | 87 | 90
  Week 32 | 0.55 (0.58) | 0.57 (0.63)
  Week 36: number analyzed (Participants) | 86 | 88
  Week 36 | 0.60 (0.60) | 0.56 (0.64)
  Week 40: number analyzed (Participants) | 84 | 88
  Week 40 | 0.55 (0.56) | 0.61 (0.67)
  Week 44: number analyzed (Participants) | 82 | 89
  Week 44 | 0.53 (0.57) | 0.58 (0.66)
  Week 48: number analyzed (Participants) | 84 | 89
  Week 48 | 0.53 (0.61) | 0.57 (0.66)
  LOCF visit | 0.55 (0.61) | 0.56 (0.66)

42. Secondary Outcome: Functional Assessment of Chronic Illness Therapy - Fatigue (FACIT-F) up to Week 24
Description: The symptom-specific measure FACIT-F assesses chronic illness therapy with special emphasis on fatigue in the past 7 days and consists of 5 dimensions: 1) physical well- being, 2) social/family well-being, 3) emotional well-being, 4) functional well-being, and 5) additional concerns. Each of the questions is categorically answered using the scales 0=not at all, 1=a little bit, 2=somewhat, 3=quite a bit, and 4=very much for a total possible FACIT-F score of 0 to 160. The figures are reversed during score calculations, so that higher score values indicate more favorable conditions.
Time Frame: From baseline to Week 24
Population: Analysis was conducted on the FAS
Measure: Mean (Standard Deviation); unit: FACIT-F score
Arm/Group | Phase 1: Tocilizumab Monotherapy | Phase 1: Combination Therapy
Number analyzed (Participants) | 74 | 327
FACIT-F score
  Baseline | 81.72 (24.75) | 89.16 (24.49)
  Week 2: number analyzed (Participants) | 74 | 319
  Week 2 | 86.64 (25.00) | 95.82 (25.42)
  Week 4: number analyzed (Participants) | 73 | 312
  Week 4 | 92.26 (25.30) | 99.54 (27.15)
  Week 8: number analyzed (Participants) | 73 | 300
  Week 8 | 96.45 (25.88) | 103.46 (27.25)
  Week 12: number analyzed (Participants) | 70 | 296
  Week 12 | 98.29 (25.47) | 104.08 (26.79)
  Week 16: number analyzed (Participants) | 69 | 292
  Week 16 | 98.41 (27.08) | 105.51 (26.94)
  Week 20: number analyzed (Participants) | 65 | 284
  Week 20 | 102.46 (27.24) | 104.91 (27.47)
  Week 24: number analyzed (Participants) | 64 | 281
  Week 24 | 104.36 (27.16) | 107.01 (27.60)
  LOCF visit | 101.38 (28.24) | 104.65 (28.07)

43. Secondary Outcome: Functional Assessment of Chronic Illness Therapy - Fatigue (FACIT-F) up to Week 48
Description: as for outcome 42
Time Frame: Baseline, from week 28 until week 48
Population: Analysis was conducted on the FAS.
Measure: Mean (Standard Deviation); unit: FACIT-F score
Arm/Group | Phase 2 Arm A1: TCZ +/- nbDMARD Once Per Week (qw) | Phase 2 Arm A2: TCZ +/- nbDMARD Every Two Weeks (q2w)
Number analyzed (Participants) | 89 | 90
FACIT-F score
  Baseline | 17.36 (5.16) | 17.13 (5.67)
  Week 28: number analyzed (Participants) | 88 | 90
  Week 28 | 23.50 (3.82) | 23.12 (4.47)
  Week 32: number analyzed (Participants) | 87 | 90
  Week 32 | 23.62 (4.16) | 22.98 (4.86)
  Week 36: number analyzed (Participants) | 86 | 88
  Week 36 | 23.23 (4.21) | 22.90 (4.64)
  Week 40: number analyzed (Participants) | 84 | 88
  Week 40 | 23.39 (4.40) | 23.02 (4.38)
  Week 44: number analyzed (Participants) | 82 | 89
  Week 44 | 23.48 (4.21) | 23.13 (4.45)
  Week 48: number analyzed (Participants) | 84 | 89
  Week 48 | 23.95 (3.79) | 22.87 (4.87)
  LOCF visit | 23.69 (4.07) | 22.88 (4.85)

ADVERSE EVENTS:
Time Frame: After initiation of study drug, all AEs, regardless of relationship to study drug, are reported until study closure.
Description: In this section the arms are not mutually exclusive because they report AE data across two different phases of the study. The patients in phase 2 groups B,C and D were considered in this study for safety reporting purposes only.
  In Non Serious Adverse events section data was calculated separately according to the two different phases of the study, i.e. Phase 1 mono-therapy and Phase 1 combination therapy groups, and the Phase 2 groups.
Arm/Group | Phase 1: Tocilizumab Monotherapy | Phase 1: Combination Therapy | Phase 2 Arm A1: TCZ +/- nbDMARD Once Per Week (qw) | Phase 2 Arm A2: TCZ +/- nbDMARD Every Two Weeks (q2w) | Phase 2 Arm B: Participants With Low Disease Activity | Phase 2 Arm C: Moderate EULAR Response at Week 24 | Phase 2 Arm D: Non Responders
All-Cause Mortality (participants affected / at risk) | 0/74 | 1/327 | 0/89 | 0/90 | 0/95 | 2/67 | 0/2
Serious Adverse Events (participants affected / at risk) | 3/74 | 10/327 | 2/89 | 1/90 | 2/95 | 5/67 | 1/2
Other Adverse Events (participants affected / at risk) | 24/74 | 119/327 | 17/89 | 25/90 | 30/95 | 23/67 | 0/2
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Phase 1: Tocilizumab Monotherapy (N=74) | Phase 1: Combination Therapy (N=327) | Phase 2 Arm A1: TCZ +/- nbDMARD Once Per Week (qw) (N=89) | Phase 2 Arm A2: TCZ +/- nbDMARD Every Two Weeks (q2w) (N=90) | Phase 2 Arm B: Participants With Low Disease Activity (N=95) | Phase 2 Arm C: Moderate EULAR Response at Week 24 (N=67) | Phase 2 Arm D: Non Responders (N=2)
Neutropenia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pericarditis (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Acute coronary syndrome (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Coronary artery disease (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Myocardial infarction (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Duodenal perforation (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Intestinal obstruction (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Ascites (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Diverticular perforation (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Ileus (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Biliary fistula (Hepatobiliary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Breast abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Abscess limb (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 2 | 0 | 0 | 0 | 0 | 0
Spinal fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Metastatic malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 0
Pyelonephritis acute (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Invasive ductal breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Urinary tract neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Thrombophlebitis (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hypertensive crisis (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Phase 1: Tocilizumab Monotherapy (N=74) | Phase 1: Combination Therapy (N=327) | Phase 2 Arm A1: TCZ +/- nbDMARD Once Per Week (qw) (N=89) | Phase 2 Arm A2: TCZ +/- nbDMARD Every Two Weeks (q2w) (N=90) | Phase 2 Arm B: Participants With Low Disease Activity (N=95) | Phase 2 Arm C: Moderate EULAR Response at Week 24 (N=67) | Phase 2 Arm D: Non Responders (N=2)
Neutropenia (Blood and lymphatic system disorders) | 4 | 18 | 1 | 5 | 3 | 2 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 4 | 9 | 0 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 1 | 18 | 0 | 0 | 0 | 0 | 0
Injection site erythema (General disorders) | 6 | 10 | 0 | 0 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 2 | 23 | 9 | 7 | 3 | 4 | 0
Urinary tract infection (Infections and infestations) | 6 | 23 | 3 | 2 | 8 | 3 | 0
Transaminases increased (Investigations) | 1 | 37 | 0 | 0 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 4 | 15 | 0 | 0 | 0 | 0 | 0
Oedema peripheral (General disorders) | 0 | 0 | 0 | 1 | 3 | 4 | 0
Nasopharyngitis (Infections and infestations) | 0 | 0 | 2 | 4 | 5 | 4 | 0
Respiratory tract infection (Infections and infestations) | 0 | 0 | 2 | 3 | 5 | 3 | 0
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2 | 3 | 6 | 3 | 0
Headache (Nervous system disorders) | 0 | 0 | 2 | 1 | 0 | 4 | 0
Hypertension (Vascular disorders) | 0 | 0 | 2 | 1 | 5 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days